CLINICAL TRIAL: NCT03921840
Title: A Personalized Behavioral Intervention for Older Adults With Musculoskeletal Pain and Sleep Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00205661; P30NR018093 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-04-19 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Sleep; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Based on the self-efficacy theory, participants in the intervention arm will receive personalized, circadian-based activity guidelines, a 2-hour in person education session, real time physical activity self-monitoring, interactive prompts, biweekly phone consultation with the research team, and financial incentives for achieving weekly physical activity goal.
  Interventions: Behavioral: ELDERFITNESS
- Control (Placebo Comparator): The control group will receive general education on physical activity for older adults and continue daily activity and healthcare routine. Participants will also receive a Go4Life program book from the National Institute on Aging.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: ELDERFITNESS — In person training: Participants will receive a 2-hour in person education session with the exercise trainer. Self-monitoring: Subjects will self-monitor subjects' level of physical activity (steps & minutes of moderate activity) using the smartwatch. The Google calendar and Fitbit apps will send messages and alerts to the subject's smartwatch that encourage subjects to achieve subjects' daily goals. If a participant has low activity for 3 consecutive days, the research assistant will call the participant to either encourage the participant to adhere to the plan or provide a modified plan after consulting the exercise trainer.
  Phone consultation: Subjects will have biweekly phone consultation with the research team members to receive guidance and adjustment on activity plans. Financial incentives: The intervention will include financial incentives. Specifically, when the daily activity goal is achieved for more than four days per week, a $5 reward will be given to subjects.
  Arms: Intervention
Other: Control — General education on physical activity for older adults and continue daily activity and healthcare routine. Participants will also receive a Go4Life program book from the National Institute on Aging.
  Arms: Control

SUMMARY:
It is well recognized that physical activity/exercise is an effective intervention to improve sleep, reduce pain and improve function in a variety of pain conditions. Traditional interventions to increase physical activity are challenging in older adults due to extensive staffing requirements and low adherence. The investigators plan to conduct a pilot trial in a cohort of older adults (without dementia) with both chronic musculoskeletal pain and nocturnal sleep complaints to test the effectiveness of a 12-week personalized behavioral intervention (compared to a control group) embedded within a smartwatch application in older adults. 27 cognitively intact elders were enrolled and randomly allocated to intervention or control group. Participants in the intervention arm received a 2-hour in person education session, and personalized, circadian-based activity guidelines, with real time physical activity self-monitoring, interactive prompts, biweekly phone consultation with the research team, and financial incentives for achieving weekly physical activity goal. The control group received general education on physical activity in older adults and continue routine daily activity for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Intact cognition
* Poor sleep quality
* Self-reported presence of pain
* Capacity for mild to moderate physical activity.

Exclusion Criteria:

* Non-ambulatory or have severely impaired mobility,
* Visual or hearing impairment that interfered with assessments, and
* An acute or a terminal illness
* Neuropathic pain

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junxin Li, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was started in July 2019 and was completed in February 2020 with 27 enrollments.
  We recruited at the geriatric clinic at the John Hopkins Bayview and community senior centers in Baltimore city.
Pre-assignment Details: 24 of the 27 enrolled participants were randomly assigned to the intervention and control groups. 3 of the 27 enrolled participants withdrew from the study before completing baseline sleep data collection and group assignment
Groups:
- Intervention: Based on the self-efficacy theory, participants in the intervention arm will receive personalized, circadian-based activity guidelines, a 2-hour in person education session, real time physical activity self-monitoring, interactive prompts, biweekly phone consultation with the research team, and financial incentives for achieving weekly physical activity goal.
  ELDERFITNESS: In person training: Participants will receive a 2-hour in person education session with the exercise trainer. Self-monitoring: Subjects will self-monitor subjects' level of physical activity (steps & minutes of moderate activity) using the smartwatch. The Google calendar and Fitbit apps will send messages and alerts to the subject's smartwatch that encourage subjects to achieve subjects' daily goals. If a participant has low activity for 3 consecutive days, the research assistant will call the participant to either encourage the participant to adhere to the plan or provide a modified plan after consulting the exercise trainer.
  Phone consultation: Subjects will have biweekly phone consultation with the research team members to receive guidance and adjustment on activity plans. Financial incentives: The intervention will include financial incentives. Specifically, when the daily activity goal is achieved for more than four days per week, a $5 reward will be given to subjects.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 12 (first enrollment) | 12
Completed | 11 | 12
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.9 (7.2) | 73.2 (7.1) | 73.0 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24
Education_Some college or higher [Count of Participants; unit: Participants] | 9 | 11 | 20
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.2 (3.3) | 30.2 (6.2) | 30.7 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Objective Sleep Duration
Description: Total sleep time (minutes) will be measured using actigraph
Time Frame: Week 1, Week 14
Population: 12 participants were assigned to the intervention group. One participant withdrew during the intervention. There were 11 participants in the invention group were included in the analysis
Measure: Mean (Standard Deviation); unit: MINUTE
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
MINUTE | 19 (41.2) | 2.5 (30.3)

2. Primary Outcome: Change in Sleep Efficiency as Assessed by Actigraphy
Description: Sleep efficiency (reported as a percentage)will be measured using actigraph
Time Frame: Week 1, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 12
percent | 5.1 (3.9) | -0.8 (8.4)

ADVERSE EVENTS:
Time Frame: during the 16 week of study participation
Description: Older adults without physical and cognitive impairment were recruited. The exercise intervention is individualized and has a minimal risk.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03921840/Prot_SAP_000.pdf